CLINICAL TRIAL: NCT00931385
Title: Characterisation of 24-hour FEV1-time Profiles of Inhaled BI 1744 CL and Inhaled Foradil Iin Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Characterization of 24 Hour Spirometry Profiles of Inhaled BI 1744 CL and Inhaled Foradil in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.24
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Formoterol Fumarate

ARMS (4):
- BI 1744 (Olodaterol) Low Dose (Experimental): BI1744 Low Dose once daily
  Interventions: Drug: bi1744
- BI 1744 (Olodaterol) Med Dose (Experimental): BI 1744 Med Dose once daily
  Interventions: Drug: BI 1744
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo
- Foradil (Active Comparator): Foradil 12 mcg twice daily
  Interventions: Drug: Foradil

INTERVENTIONS:
Drug: BI 1744 — BI1744 Respimat Med Dose Once Daily
  Arms: BI 1744 (Olodaterol) Med Dose
Drug: bi1744 — 1744 low dose
  Arms: BI 1744 (Olodaterol) Low Dose
Drug: Placebo — Placebo Respimat and Foradil Placebo
  Arms: Placebo
Drug: Foradil — Foradil 12 mcg twice daily and Placebo Respimat
  Arms: Foradil

SUMMARY:
The study is intended to characterize the lung function profile of BI1744 in COPD patients where patients will perform pulmonary function tests at regular intervals for 24 hours at the end of a 6 week treatment period. Each patient will receive all four treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate with confirmed diagnosis of COPD
* 40 years of age or older
* having a 10 pack year smoking history
* able to perform serial pulmonary function tests
* able to use both a DPI and Respimat device

Exclusion Criteria:

* Significant other disease
* clinically relevant abnormal hematology, chemistry, or urinalysis
* history of asthma
* diagnosis of thyrotoxicosis
* paroxysmal tachycardia related to beta agonists
* history of MI within 1 year, cardiac arrhythmia, hospitalization for heart failure within 1 year
* active tuberculosis, cystic fibrosis, clinically evident bronchiectasis
* significant alcohol or drug use
* pulmonary resection
* taking oral beta adrenergics
* taking unstable oral steroids
* daytime oxygen
* enrolled in rehabilitation program
* enrolled in another study or taking investigational products
* pregnant or nursing women, women of child bearing potential not willing to use two methods of birth control
* those who are not willing to comply with pulmonary medication washouts

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- United States (11):
  - 1222.24.24011 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1222.24.24009 Boehringer Ingelheim Investigational Site, Overland Park, Kansas
  - 1222.24.24007 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1222.24.24002 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1222.24.24010 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1222.24.24004 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1222.24.24006 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1222.24.24005 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.24.24008 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.24.24001 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.24.24003 Boehringer Ingelheim Investigational Site, Union, South Carolina

REFERENCES:
- [Derived] Feldman GJ, Bernstein JA, Hamilton A, Nivens MC, Korducki L, LaForce C. The 24-h FEV1 time profile of olodaterol once daily via Respimat(R) and formoterol twice daily via Aerolizer(R) in patients with GOLD 2-4 COPD: results from two 6-week crossover studies. Springerplus. 2014 Aug 9;3:419. doi: 10.1186/2193-1801-3-419. eCollection 2014. PMID 25187881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, double-dummy, placebo-controlled, 4-way crossover trial. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Groups:
- Olo 5mcg / Foradil 12mcg / Placebo / Olo 10mcg: Patients were administered Olodaterol 5 mcg qd in the first period, Foradil 12 mcg bid in the second period, matching Placebo in the third period and Olodaterol 10 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Foradil 12mcg / Olo 10mcg / Olo 5mcg / Placebo: Patients were administered Foradil 12 mcg bid in the first period, Olodaterol 10 mcg qd in the second period, Olodaterol 5 mcg qd in the third period and matching Placebo in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Olo 10mcg / Placebo / Foradil 12mcg / Olo 5mcg: Patients were administered Olodaterol 10 mcg qd in the first period, matching Placebo in the second period, Foradil 12 mcg bid in the third period and Olodaterol 5 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
- Placebo / Olo 5mcg / Olo 10mcg / Foradil 12mcg: Patients were administered matching Placebo in the first period, Olodaterol 5 mcg qd in the second period, Olodaterol 10 mcg qd in the third period and Foradil 12 mcg bid in the fourth period. Olodaterol was administered via the Respimat inhaler, Foradil was administered via the Aerolizer inhaler.
Period: Overall Study
Arm/Group | Olo 5mcg / Foradil 12mcg / Placebo / Olo 10mcg | Foradil 12mcg / Olo 10mcg / Olo 5mcg / Placebo | Olo 10mcg / Placebo / Foradil 12mcg / Olo 5mcg | Placebo / Olo 5mcg / Olo 10mcg / Foradil 12mcg
Started | 25 | 23 | 25 | 26
Completed | 23 | 21 | 24 | 21
Not Completed | 2 | 2 | 1 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set, i.e., all treated patients.
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. 99 patients were assigned randomly to one of 4 treatment sequences in which they received each of 4 treatments, two doses (5 microgram (mcg) or 10 mcg) of Olodaterol (Olo) once daily (qd) delivered via the Respimat inhaler or Foradil (Form) 12 mcg twice daily (bid) delivered via the Aerolizer inhaler or equivalent placebo delivered by Respimat Inhaler or Aerolizer Inhaler. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of treatment (baseline) and -30 min (zero time), 30 min, 60 min, 2 hour (h) , 3 h, 4 h, 6 h, 8 h, 10 h, 11 h 50 min relative to am dose after six weeks of treatment
Population: Full analysis set (FAS). FAS is defined as all patients with the baseline (pre-dose) data and any evaluable post-dosing data for the first co-primary endpoint FEV1AUC 0-12h.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler or Aerolizer Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg Bid: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.060 (0.020) | 0.088 (0.021) | 0.088 (0.021) | 0.081 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with center, treatment and period as fixed effects and patients within center as random effect; Mean Difference (Final Values) = 0.148, 95% CI [0.113 to 0.183], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.148, 95% CI [0.113 to 0.183], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.106 to 0.177], Standard Error of Mean 0.018 — Form 12 mcg bid minus Placebo

2. Primary Outcome: FEV1 Area Under Curve 12-24h (AUC 12-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit, just prior to administration of the morning dose of randomized treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of treatment (baseline) and 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat resp. Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.123 (0.021) | -0.014 (0.022) | 0.004 (0.022) | 0.049 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.109, 95% CI [0.073 to 0.146], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.127, 95% CI [0.091 to 0.164], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.135 to 0.209], Standard Error of Mean 0.019 — Form 12 mcg bid minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 h (AUC 0-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 h and 10 min prior to am dose on the first day of treatment (baseline) and -30 min, 30 min, 60 min, 2h, 3h, 4h, 6h, 8h, 10h, 11 hr 50 min,12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment.
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.092 (0.020) | 0.037 (0.021) | 0.046 (0.021) | 0.065 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.094 to 0.163], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.137, 95% CI [0.103 to 0.172], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.122 to 0.191], Standard Error of Mean 0.018 — Form 12 mcg bid minus Placebo

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FEV1 AUC 0-3h was calculated from 0-3hours post-dose using the trapezoidal rule, divided by the observation time (3 h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to the last am dose after six weeks of treatment
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.030 (0.020) | 0.134 (0.021) | 0.135 (0.021) | 0.168 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.126 to 0.201], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.127 to 0.202], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.198, 95% CI [0.160 to 0.236], Standard Error of Mean 0.019 — Form 12 mcg bid minus Placebo

5. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values at the randomisation visit. Peak (0-3h) values were obtained within 0 - 3 hours after the last am dose after six weeks of treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | 0.034 (0.022) | 0.208 (0.022) | 0.200 (0.022) | 0.251 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.135 to 0.214], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.166, 95% CI [0.127 to 0.206], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.218, 95% CI [0.178 to 0.257], Standard Error of Mean 0.020 — Form 12 mcg bid minus Placebo

6. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline trough FEV1 was defined as the mean of the available pre-dose trough FEV1 values at the randomisation visit. Trough values were obtained 30 minutes prior to the last am dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.093 (0.023) | 0.012 (0.024) | 0.020 (0.024) | 0.040 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.106, 95% CI [0.064 to 0.147], Standard Error of Mean 0.021 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.113, 95% CI [0.072 to 0.155], Standard Error of Mean 0.021 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.133, 95% CI [0.092 to 0.175], Standard Error of Mean 0.021 — Form 12 mcg bid minus Placebo

7. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 1
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.086 (0.036) | 0.139 (0.036) | 0.142 (0.036) | 0.117 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.226, 95% CI [0.167 to 0.284], Standard Error of Mean 0.030 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 95% CI [0.170 to 0.287], Standard Error of Mean 0.030 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.203, 95% CI [0.144 to 0.262], Standard Error of Mean 0.030 — Form 12 mcg bid minus Placebo

8. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 2
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.164 (0.036) | -0.016 (0.037) | 0.008 (0.037) | 0.088 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.087 to 0.207], Standard Error of Mean 0.030 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.171, 95% CI [0.112 to 0.231], Standard Error of Mean 0.030 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.251, 95% CI [0.191 to 0.311], Standard Error of Mean 0.030 — Form 12 mcg bid minus Placebo

9. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 3
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.125 (0.035) | 0.061 (0.035) | 0.075 (0.035) | 0.102 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.186, 95% CI [0.132 to 0.241], Standard Error of Mean 0.028 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.200, 95% CI [0.145 to 0.254], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.227, 95% CI [0.172 to 0.282], Standard Error of Mean 0.028 — Form 12 mcg bid minus Placebo

10. Secondary Outcome: Peak FVC (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FVC was defined as the mean of the available pre-dose peak FVC values at the randomisation visit. Peak FVC (0-3h) was obtained within 0 - 3 hours after the last am dose of study drug after 6 weeks of treatment. Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | 0.107 (0.038) | 0.368 (0.039) | 0.360 (0.039) | 0.410 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.261, 95% CI [0.191 to 0.330], Standard Error of Mean 0.035 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.252, 95% CI [0.183 to 0.322], Standard Error of Mean 0.036 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.302, 95% CI [0.232 to 0.372], Standard Error of Mean 0.036 — Form 12 mcg bid minus Placebo

11. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline trough FVC was defined as the mean of the available pre-dose trough FVC values at the randomisation visit. Trough values were obtained 30 minutes prior to the last am dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with center, treatment and period as fixed effects and patient within center as random.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Form 12 mcg Bid
Number analyzed (Participants) | 93 | 92 | 91 | 90
Liter | -0.117 (0.039) | 0.037 (0.040) | 0.037 (0.040) | 0.066 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.154, 95% CI [0.087 to 0.221], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.154, 95% CI [0.086 to 0.221], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Form 12 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.183, 95% CI [0.115 to 0.250], Standard Error of Mean 0.034 — Form 12 mcg bid minus Placebo

12. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 6 weeks
Population: Treated set.
Measure: Number; unit: participants
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Form 12 mcg: Foradil 12 mcg bid (morning and evening) delivered by the Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Form 12 mcg
Number analyzed (Participants) | 96 | 95 | 92 | 93
participants
  Heart rate increased | 0 | 1 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Form 12 mcg
Serious Adverse Events (participants affected / at risk) | 4/96 | 4/95 | 2/92 | 1/93
Other Adverse Events (participants affected / at risk) | 5/96 | 4/95 | 1/92 | 3/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=96) | Olo 5 mcg (N=95) | Olo 10 mcg (N=92) | Form 12 mcg (N=93)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=96) | Olo 5 mcg (N=95) | Olo 10 mcg (N=92) | Form 12 mcg (N=93)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication